CLINICAL TRIAL: NCT06957522
Title: Comparison of the Effectiveness of Face to Face Rehabilitation and Telerehabilitation in Infants With Congenital Muscular Torticollis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gökçen Erol, MSc Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GErol1
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Infant; Torticollis Congenital; Neurodevelopment Treatment; Telerehabilitation; Physiotherapy and Rehabilitation
Keywords: telerehabilitation; congenital torticollis; infant; neurodevelopment treatment; physiotherapy and rehabilitation
MeSH Terms: conditions — Congenital torticollis | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: The study will compare the effectiveness of face-to-face and telerehabilitation methods in infants diagnosed with congenital muscular torticollis aged 0-6 months. The sample size was determined as 42 by preliminary analysis. Infants diagnosed with congenital muscular torticollis aged 0-6 months, who meet the inclusion criteria and whose parents volunteer to participate in the exercise program will be included in the study. Infants whose parents sign the informed consent form will be included in the study. Participants will be divided equally into two groups (face-to-face rehabilitation group and telerehabilitation group) (n=21) by simple randomization method. Treatment will be applied to both groups for 8 weeks, 2 days a week and each session will be 30 minutes. The treatment content includes exercises to increase active neck range of motion, activities supporting symmetrical movements, family education, home program and practices supporting gross motor development.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): The telerehabilitation group receives the same structured, neurodevelopmentally-based rehabilitation program as the face-to-face group. However, the delivery method-via online video conferencing (Zoom)-represents a novel mode of application for this specific intervention in infants with congenital muscular torticollis (CMT).
  To date, this therapeutic program has not been delivered through telehealth for this population, and its feasibility, effectiveness, and comparability to the conventional face-to-face method have not yet been studied. Therefore, this arm is considered experimental as it involves a new and previously untested method of intervention delivery, even though the therapeutic content remains the same.
  Interventions: Other: telerehabilitation
- Face to face rehabilitation (Active Comparator): The face-to-face rehabilitation group receives a structured, neurodevelopmental treatment program that is already in routine clinical use for infants with congenital muscular torticollis (CMT). It represents the current standard method of delivering this intervention in clinical settings.
  Since the objective of the study is to compare the effectiveness of a novel telerehabilitation delivery model against this established, routinely used face-to-face method, the face-to-face arm serves as the active comparator. This arm provides a baseline for evaluating the outcomes of the experimental telerehabilitation approach.
  Interventions: Other: face to face rehabilitation

INTERVENTIONS:
Other: face to face rehabilitation — The face-to-face rehabilitation program will be delivered in a clinical setting to infants aged 0-6 months with congenital muscular torticollis (CMT). It is based on neurodevelopmental treatment (NDT) principles and consists of:
  Passive range of motion (ROM) exercises for the neck
  Active ROM exercises for the neck and trunk
  Activities to promote the development of symmetrical movement
  Environmental modification suggestions for the home setting
  Parent/caregiver education and training
  Sessions will be conducted twice per week, 30 minutes per session, over a total of 8 weeks.
  In addition, an individualized home exercise program will be prescribed for each infant based on their specific needs. Frequency and duration of the home exercises may vary accordingly.
  Arms: Face to face rehabilitation
Other: telerehabilitation — The telerehabilitation program provides the same therapeutic content as the face-to-face rehabilitation group but will be delivered remotely via the Zoom video conferencing platform. The program will be applied to infants aged 0-6 months with congenital muscular torticollis (CMT) and is based on neurodevelopmental treatment (NDT) principles, including:
  Passive range of motion (ROM) exercises for the neck
  Active ROM exercises for the neck and trunk
  Activities for symmetrical movement development
  Environmental modification suggestions
  Parent/caregiver education and guidance
  Sessions will be conducted via live video calls, twice per week, 30 minutes per session, for 8 weeks.
  Each family will also receive an individualized home exercise program, with its frequency and duration adapted to the infant's needs.
  Arms: Telerehabilitation

SUMMARY:
Who is this study for? This study is designed for infants aged 0-6 months who have been diagnosed with Congenital Muscular Torticollis (CMT). CMT is a condition observed at birth or shortly after, characterized by the shortening of the sternocleidomastoid (SCM) muscle, leading to the baby's head tilting to one side and rotating to the opposite side. It affects both boys and girls and may result in limited neck movement, abnormal posture, facial asymmetry, and potential developmental delays if left untreated.

What is the purpose of this study? The goal of this study is to compare the effectiveness of two different physical therapy methods-face-to-face rehabilitation and telerehabilitation-in treating infants with CMT. In addition to evaluating the outcomes of these two therapy methods, this research also aims to provide families with reliable, accessible information through a web-based educational platform.

Why is this study important? Early diagnosis and intervention are crucial for optimal recovery in infants with CMT. Studies show that infants who begin therapy by one month of age have up to a 98% chance of full recovery. However, if diagnosis and treatment are delayed, the recovery process can take longer and may be less effective. This study will help determine if online (telerehabilitation) sessions can be just as effective as traditional face-to-face therapy, offering a flexible and accessible treatment option for families.

What are the benefits of participating?

* Access to a structured, evidence-based rehabilitation program for your child
* Guidance from trained pediatric physiotherapists
* Increased awareness and knowledge about CMT through a web-based family education platform
* Contribution to research that may benefit other children and families in the future
* Evaluation of your baby's progress through professional assessments

What will the therapy program involve?

Participants will be randomly assigned to either a face-to-face or telerehabilitation group. Both groups will follow the same therapy program, focusing on:

* Increasing passive and active neck movements
* Promoting symmetrical head and body movement
* Providing recommendations for environmental adjustments
* Educating parents or caregivers on home-based exercises and care

Program structure:

* Face-to-face group: Therapy sessions will be conducted in a clinic setting, twice a week for 30 minutes each session, over a period of 8 weeks.
* Telerehabilitation group: Therapy sessions will be conducted via Zoom, with the same frequency, duration, and content as the face-to-face sessions.

How will outcomes be measured?

Infants will be assessed before and after the 8-week therapy period for:

* Passive cervical range of motion (rotation and lateral flexion)
* Gross motor function
* Muscle function Parental adherence to the home program will also be evaluated through a questionnaire. A follow-up will be conducted one month after therapy ends.

How can I participate? If your infant is aged 0-6 months and has been diagnosed with CMT, you may be eligible to participate. You will need access to a device with internet for telerehabilitation sessions, if assigned to that group. Participation is voluntary and free of charge. Families will receive detailed instructions and ongoing support throughout the program.

Additional Resources:

As part of this study, a web-based educational platform will be made available to all participating families. This platform will include:

* Clear explanations about CMT
* Instructional videos and home exercise guides
* Tips for daily care and positioning
* Frequently asked questions (FAQ) for parents Why is this research unique? This is one of the first studies to scientifically compare face-to-face and online rehabilitation for CMT infants, while also providing a reliable online resource for families. It aims to help develop alternative, flexible care models that meet the diverse needs of families and infants.

Contact Information:

If you are interested in participating or would like more information, please contact our research team at:

[fgokcenalaca@gmail.com / +905534646606] We are committed to supporting your child's health and development. Thank you for considering being a part of this important study.

DETAILED DESCRIPTION:
Study Design This study is designed as a prospective, randomized controlled clinical trial to compare the effectiveness of face-to-face and telerehabilitation programs in infants diagnosed with Congenital Muscular Torticollis (CMT) between 0-6 months of age. Both groups will receive an identical intervention protocol, consisting of two sessions per week, 30 minutes each, over a total of 8 weeks.

The intervention content includes exercises to increase active cervical range of motion (ROM), activities promoting symmetrical movements, family education, home exercise programs, and practices to support gross motor development.

Study Population and Sample Size In a study by Lee et al. (2015), the effect size for head tilt angle was calculated as 1.45. Based on this effect size, with α = 0.05 and a power of 99%, the required sample size was determined to be 19 participants per group. With an anticipated 15% drop-out rate, the total sample size was set at 42 infants.

Inclusion Criteria

* Diagnosed with Congenital Muscular Torticollis (CMT)
* Infants under 6 months of age
* Classified as level 1 to 3 according to the CMT classification system

Exclusion Criteria

* Presence of ocular torticollis
* Neurological complications (e.g., cerebral palsy)
* Congenital anomalies of the cervical spine or spinal cord
* Visual or auditory impairments

Participant Recruitment and Randomization Infants referred with a diagnosis of CMT will be screened, and those who meet the inclusion criteria will be invited to participate. Families will be informed in detail, and written informed consent will be obtained. Participants will be randomly allocated into two groups (face-to-face and telerehabilitation) using computer-generated simple randomization (n = 21 per group).

Outcome Measures

All outcomes will be assessed at baseline and after the 8-week intervention period:

* Passive cervical range of motion (ROM): Measured using a goniometer
* Alberta Infant Motor Scale (AIMS): To evaluate gross motor development
* Head tilt angle: Assessed using a standardized photographic measurement protocol
* Muscle Function Scale: To assess the functional status of neck muscles
* Adherence to home exercise program: Evaluated through a parent-reported checklist

Statistical Analysis Data will be analyzed using SPSS version 26.0 (IBM Corp, Armonk, NY). Descriptive statistics (mean, standard deviation, frequency, percentage) will be presented for both categorical and continuous variables. The Levene test will be used to assess homogeneity of variances. For between-group comparisons, independent-samples t-test will be used for normally distributed data; otherwise, the Mann-Whitney U test will be applied. A p-value < 0.05 will be considered statistically significant.

Research Hypotheses H₀: There is no significant difference between telerehabilitation and face-to-face rehabilitation in infants with CMT in terms of cervical ROM, gross motor function, muscle function, and parental adherence.

H₁: There is a significant difference between telerehabilitation and face-to-face rehabilitation in infants with CMT in terms of cervical ROM, gross motor function, muscle function, and parental adherence.

ELIGIBILITY:
Inclusion Criteria:

* Infants aged 0 to 6 months
* Diagnosed with congenital muscular torticollis (CMT)
* Classified as Grade 1 to 3 CMT severity based on clinical assessment

Exclusion Criteria:

* Plagiocephaly
* Ocular torticollis
* Neurological complications
* Musculoskeletal disorders of the cervical spine
* Visual impairments
* Hearing impairments

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Passive Cervical Range of Motion (Lateral Flexion and Rotation) | Baseline, Week 8 (post-treatment), and 1-month follow-up
  Passive range of motion (ROM) of the neck, specifically lateral flexion and rotation, will be assessed using an arthrodial goniometer. Measurements will be taken at three time points:
  Baseline (Pre-intervention) Post-intervention (At the end of 8 weeks of rehabilitation) Follow-up (1 month after the end of the intervention) This outcome aims to evaluate changes in cervical mobility in response to the rehabilitation programs.
Head Tilt Angle (Still Photography Method) | Baseline, Week 8 (post-treatment), and 1-month follow-up
  Head tilt will be assessed using the Still Photography Method, a standardized photographic procedure:
  A photograph of the infant is taken in a supin position. A horizontal line is drawn connecting the pupils of both eyes (inter-pupillary line).
  A second line is drawn connecting the acromion processes of both shoulders. The acute angle between these two lines is measured to quantify the degree of head tilt.
  This method allows for an objective and reliable evaluation of head posture asymmetry in infants with congenital muscular torticollis (CMT).

SECONDARY OUTCOMES:
Muscle Function Test (MFT) | Baseline, Week 8 (post-treatment), and 1-month follow-up
  The Muscle Function Test (MFT) is a visual assessment tool used to evaluate the infant's head-righting response. The procedure is performed as follows:
  The infant is held in a vertical position, facing a mirror.
  The infant is then slowly moved into a horizontal position, toward the side of the shortened sternocleidomastoid (SCM) muscle.
  The evaluator observes the head and neck righting reaction, focusing on the infant's ability to align the head vertically in response to the positional change.
  The test is scored on a 6-point scale (0-5) based on the alignment of the head relative to the vertical axis.
Alberta Infant Motor Scale (AIMS) | Baseline, Week 8 (post-treatment), and 1-month follow-up
  The Alberta Infant Motor Scale (AIMS) will be used to assess gross motor development in infants. AIMS is a standardized observational assessment tool designed to evaluate motor performance and monitor the effectiveness of early interventions in infants aged 0 to 18 months.
  The test consists of 58 items and takes approximately 10 minutes to administer. The infant's spontaneous movements are observed in four positions: supine, prone, sitting, and standing, without any physical contact.
  Each item that the infant successfully performs is scored as 1 point. The total raw score is then converted into a percentile score based on age norms. The percentile rank reflects the infant's motor performance in comparison to age-matched peers.
  According to the normative chart:
  Percentiles of 5% or below indicate atypical development.
  Percentiles below 10% suggest the infant is at risk for motor delay.
  Scores are categorized as normal, suspicious, or abnormal.
  The AIMS has demonstrated strong va

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Study Director — Istanbul University-Cerrahpasa,Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Division of Physiotherapy and Rehabilitation; GÖKÇEN EROL, Principal Investigator — Istanbul University-Cerrahpasa, Graduate School of Health Sciences
Locations (1):
- Istanbul University - Cerrahpasa, Faculty of Health Sciences, Büyükçekmece Campus, Alkent 2000 Mah. Yiğittürk Street No:5/9/1, Büyükçekmece/Istanbul, Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Result] Rodriguez-Huguet M, Rodriguez-Almagro D, Rosety-Rodriguez MA, Vinolo-Gil MJ, Ayala-Martinez C, Gongora-Rodriguez J. Effectiveness of the Treatment of Physiotherapy in the Congenital Muscular Torticollis: A Systematic Review. Children (Basel). 2023 Dec 20;11(1):8. doi: 10.3390/children11010008. PMID 38275429
- [Result] Sargent B, Coulter C, Cannoy J, Kaplan SL. Physical Therapy Management of Congenital Muscular Torticollis: A 2024 Evidence-Based Clinical Practice Guideline From the American Physical Therapy Association Academy of Pediatric Physical Therapy. Pediatr Phys Ther. 2024 Oct 1;36(4):370-421. doi: 10.1097/PEP.0000000000001114. Epub 2024 Oct 1. PMID 39356257
- [Result] Castilla A, Gonzalez M, Kysh L, Sargent B. Informing the Physical Therapy Management of Congenital Muscular Torticollis Clinical Practice Guideline: A Systematic Review. Pediatr Phys Ther. 2023 Apr 1;35(2):190-200. doi: 10.1097/PEP.0000000000000993. Epub 2023 Jan 10. PMID 36637442
- [Result] Kaplan SL, Coulter C, Sargent B. Physical Therapy Management of Congenital Muscular Torticollis: A 2018 Evidence-Based Clinical Practice Guideline From the APTA Academy of Pediatric Physical Therapy. Pediatr Phys Ther. 2018 Oct;30(4):240-290. doi: 10.1097/PEP.0000000000000544. PMID 30277962